CLINICAL TRIAL: NCT05540158
Title: A Mobile Integrated Health Intervention for the Management of Acute-phase Exacerbation of Congestive Health Failure and Chronic Obstructive Pulmonary Disease
Brief Title: A Mobile Integrated Health Intervention to Manage Congestive Health Failure and Chronic Obstructive Pulmonary Disease
Status: Withdrawn | Type: Observational
Why Stopped: The study design underwent substantial modifications, including changes to the population, intervention, and primary outcomes. As a result, a new trial was registered under a separate ClinicalTrials.gov identifier (NCT06000696).
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Laurel O'Connor, Assistant Professor, University of Massachusetts, Worcester
Other Study IDs: STUDY00000126
Record Dates: First submitted 2022-09-10; First posted 2022-09-14 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Congestive Heart Failure; Copd
Keywords: Allied Health Personnel; Mobile Health Units; Delivery of Health Care, Integrated
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Mobile Integrated Health Intervention — Subjects will have access to "on-demand" mobile integrated health program for acute symptoms. Subjects will be educated on the nature and capabilities of the MIH community paramedics and will be able to call a hotline for unscheduled visits 24 hours a day, 7 days a week if they wish to be evaluated for acute symptoms or changes in their condition. All visits entail focused history and physical exam with community paramedic, portable diagnostics as indicated, and telehealth visit with a physician

SUMMARY:
Episodic and disjointed medical care for older, community-dwelling adults with chronic obstructive pulmonary disease (COPD) and congestive heart failure (CHF) leave them vulnerable to adverse events such as worsening disease trajectories, frequent emergency department (ED) utilization, and avoidable hospital admissions. It is imperative that an alternative means of health delivery be developed, establishing a coordinated, flexible care model to connect patients with the appropriate resources to address their acute needs and integrate with their medical homes to navigate fraught moments in their disease management.

The Mobile integrated health (MIH) care delivery model may offer a solution by providing flexible and innovative on-demand care in the comfort of patients' homes. The MIH paradigm expands the use of highly trained paramedics outside of their traditional EMS role, by dispatching them into the community to perform in-home medical evaluations and treatment(s) in consultation with an actively involved, remotely located, supervising physician. These "community paramedics" evaluate patients and render care using mobile diagnostics and a variety of medications, allowing patients to remain in place until they can be evaluated definitively on an ambulatory basis.

Utilizing a model of on-demand community paramedic visits paired with a telehealth consultation with a physician, this intervention will manage patients in place until they can access planned ambulatory follow up, decreasing the use of prehospital emergency transport services, emergency department utilizations, and hospital admissions as well as limiting transitions of care and allowing ambulatory providers to maintain longitudinal oversight of disease management

The objective of this project is to study the feasibility of the refined MIH model for the care of community dwelling patients with congestive heart failure and chronic obstructive pulmonary disease. Investigators will conduct a small pre/post pilot intervention trial enrolling 50 patients into a pilot MIH program. Primary outcomes will include participant satisfaction, patient activation, and subject retention. Investigators will also collect outcomes data including ED visits, hospitalizations, and hospital lengths of stay.

ELIGIBILITY:
Inclusion Criteria:

* Community Dwelling
* Residing in the catchment area of Worcester and Shrewsbury Massachusetts
* member of the UMMHC accountable care organization for at least one year prior to the implementation of the intervention
* Carry a diagnosis of congestive heart failure or chronic obstructive pulmonary disease
* Adult over eighteen
* Fluent in English
* Able to participate in a verbal interview either in-person or via zoom video conference
* Able to provide informed consent to participate in the study

Exclusion Criteria:

* Adults unable to consent
* Non-English-speaking adults
* Prisoners
* Patients under age 18 years
* Trainees, including medical students, resident physicians, and fellows will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community dwelling adults in Worcester county Massachusetts who are members of the Umass Memorial accountable care organization who have a diagnosis of chronic obstructive pulmonary disease or congestive heart failure
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Subject retention in study | 1 year after initial recruitment
  The number of subjects who participate in study for entire 1 year duration
Subject reported acceptability of the MIH program | baseline, 6 months and 1 year after initial recruitment
  Subjects will self report their satisfaction and utilization history with MIH program using 5 point Likert scales (5-Strongly Agree, 4-Agree, 3-Neutral, 2-Disagree, 1-Strongly Disagree) evaluating their experiences with the MIH service. A high score indicates greater satisfaction
Patient activation measure | baseline, 6 months and 1 year after initial recruitment
  Measure of a subject's knowledge, skills and confidence to manage their own health and well-being. Questions are answered on the following scale: (5-Strongly Agree, 4-Agree, 3-Neutral, 2-Disagree, 1-Strongly Disagree). A higher score indicates greater patient activation.
Brief Illness Perception Questionnaire | baseline, 6 months and 1 year after initial recruitment
  Measures subject's self-reported perception of their chronic illness through several statements that patients agree with on a 1-10 scale, with 10 being most strongly agree.
Patient satisfaction questionnaire | baseline, 6 months and 1 year after initial recruitment
  Measures subject's self-reported satisfaction with their health care. Questions are answered on the following scale: (5-Strongly Agree, 4-Agree, 3-Neutral, 2-Disagree, 1-Strongly Disagree). A higher score indicates greater patient satisfaction.

SECONDARY OUTCOMES:
Healthcare Utilizations | 1 year prior to, and 6 months and 1 year after initial recruitment
  number of MIH, ambulatory, and emergency services utilizations

IPD SHARING:
Plan to Share IPD: Undecided